CLINICAL TRIAL: NCT01706484
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Parallel Group Trial to Assess Efficacy and Safety of Two Dosages of a Herbal Medicinal Product (Dry Extract BNO 1016) in Patients With Chronic Rhinosinusitis
Brief Title: Efficacy and Safety of Two Dosages of a Herbal Medicinal Product (Dry Extract BNO 1016) in Chronic Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRS-02; 2011-003623-35 (EudraCT Number)
Record Dates: First submitted 2012-09-04; First posted 2012-10-15 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Sinusitis
Keywords: randomized clinical trial; chronic rhinosinusitis; herbal extract BNO 1016; exacerbation; pharmacoeconomic; quality of life
MeSH Terms: interventions — BNO 1016; Plant Extracts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 80 mg BNO 1016 und placebo (Experimental): 2 tablets (one containing 80 mg BNO 1016 and one placebo) by mouth 3 times daily
  Interventions: Drug: BNO 1016
- 160 mg BNO 1016 (Experimental): 2 tablets (each containing 80 mg BNO 1016) by mouth 3 times daily
  Interventions: Drug: BNO 1016
- placebo (Placebo Comparator): 2 tablets (each without BNO 1016) by mouth 3 times daily
  Interventions: Drug: BNO 1016

INTERVENTIONS:
Drug: BNO 1016 — comparison of different dosages of drug and placebo
  Other Names: herbal plant extract,; sinupret extract mite

SUMMARY:
The purpose of this trial is to determine whether 2 different dosages of a herbal extract (240 and 480 mg/day) are more effective than placebo in the treatment of patients with chronic rhinosinusitis (average reduction of investigator's Major Symptom Score over Visit 5 and Visit 6.

DETAILED DESCRIPTION:
The clinical trial population consists of patients presenting with two or more typical symptoms of CRS and duration of symptoms of at least ≥12 weeks. The diagnosis should have been confirmed with the initial diagnosis of CRS by nasal endoscopy and/or computer tomography (CT) and by obligatory nasal endoscopy including exclusion of nasal polyps during screening phase.

A total of 885 patients will be included in this clinical trial, which will last for approximately 12 months, including screening, treatment and medication-free follow-up period as well as final reporting. The duration for the individual patient is approximately 22 weeks (Visit 1 - Visit 7). After a 2-week screening phase, treatment will be started by application of either 240 mg or 480 mg daily dose (t.i.d.) or placebo for 12 weeks followed by a medication-free follow-up period.

Symptoms often do not correlate to the findings in nasal endoscopy or CT. Therefore, efficacy in this clinical trial is defined as per clinical definition using five individual rhinosinusitis symptoms (MSS)graded by the investigator using increasing severity grading(0 = absent [none / not present], 1 = mild, 2 = moderate, 3 = severe).

Secondary outcome measures include

* single rhinosinusitis symptoms of CRS (MSSINV and MSSPAT),
* Work Productivity and Activity Impairment patient questionnaire related to General Health [WPAI:GH],
* total symptom severity by Visual Analogue Scale
* response to treatment rated by investigator and patient
* 20-Question Sino-Nasal Outcome Test [SNOT-20, only Germany]
* percentage of patients with permitted concomitant medication for the treatment of CRS
* premature termination due to exacerbations of symptoms
* post treatment course of CRS will
* pharmacoeconomic assessments
* safety and tolerability of trial treatment

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent including data protection declaration
* Male and female outpatients aged ≥18 and ≤75 years
* Diagnosis of bilateral chronic rhinosinusitis without nasal polyps confirmed by:

  * nasal endoscopy during the screening period (nasal endoscopy results not older than 2 month will be accepted) to confirm inflammation, mucopurulent discharge and/or oedema/mucosal obstruction primarily in middle meatus without nasal polyps being present
  * at the discretion of the investigator a historic CT (before screening and not older than 24 months) will be considered additionally for confirmation of bilateral involvement of middle meatus and paranasal sinuses without resolution of symptoms (mucosal changes within the ostiomeatal complex and/or sinuses)
* Bilateral chronic rhinosinusitis characterized by (V1 and V2):

  * presence of chronic rhinosinusitis symptoms for at least 12 weeks without complete resolution of symptoms prior to enrolment (V1)
  * a MSS ≥6 points and ≤12 points for each of the screening days observed by diary entries (MSSPAT)and on the days of Visit 1 and 2 (MSSINV)
  * on 5 random days of the screening period (or at least at days -5 to -1) assessed by MSSPAT and on the day of Visit 1 and 2 assessed by MSSINV: rhinorrhoea (anterior or posterior) and pain (facial pain or headache) of at least moderate intensity (score ≥2).

Exclusion Criteria:

* Sinus surgery within the last 2 years (solitary sinus puncture is allowed)
* Nasal concha surgery within the last 3 months
* Presence or history of uni- or bilateral nasal polyps
* Presence of moderate to severe co-morbid asthma, including allergic asthma
* Patients with mild asthma having exacerbations within 30 days prior to trial inclusion
* Patients with cystic fibrosis
* Patients with a positive skin prick test at V1 against allergens to which the patient might be exposed to during the expected individual trial duration, if clinically relevant (results not older than 12 months will be accepted)
* Clinically relevant perennial (e.g. patients with actual clinical symptoms of allergic rhinitis against house dust/-mite antigen) or actual seasonal allergic rhinitis
* Rhinitis medicamentosa (drug induced rhinitis)
* Aspirin-Exacerbated Respiratory Disease [AERD] (Aspirin sensitivity)
* Dentogenic sinusitis or otherwise unilateral sinusitis
* Presence of anatomical deviations of the nasal septum that significantly impair nasal and paranasal ventilation / airflow
* Known hypersensitivity to trial medication or excipients
* Patients with rare hereditary problems of fructose intolerance, galactose intolerance, lactase deficiency or glucose-galactose malabsorption or sucrase-isomaltase insufficiency
* Signs or symptoms of acute bacterial sinusitis (e.g. fever > 38.5°C, orbital complications,severe unilateral frontal headache or toothache)
* Treatment with systemic or nasal antibiotics or corticosteroids within the last 4 weeks prior to V1
* Treatment with decongestant preparations (α-sympathomimetics), analgesics (including systemic Non-Steroidal Inflammatory Drugs [NSAIDs], except paracetamol), mucolytics / secretolytics, antihistamines, or alternative medicine preparations for treatment of common cold like symptoms or with immunomodulating properties within the last 7 days prior to V1
* Patients with gastric or duodenal ulcer
* Other diseases within 5 years prior to V1, which in the opinion of the investigator disqualifies the patient for trial enrolment (e.g. liver or kidney disease, severe somatopathic, neurological and /or psychiatric diseases, history of malignancy or alcohol or drug abuse or immunodeficiency).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Average of investigator's Major Symptom Score ratings [score points] at V5 and V6 | 4 weeks
  The primary efficacy endpoint is defined as the average of investigator's Major Symptom Score ratings [score points] at V5 and V6 (arithmetic mean of 2 ratings).

SECONDARY OUTCOMES:
Patient´s MSS ratings [score points] from V5 to V6 | 4 weeks
  Arithmetic mean of approximately 28 ratings, Diary data
Investigtor´s MSS ratings [score points] at V3 | Day 8
  CRF data
Investigator´s MSS ratings [score points] at V4 | Day 29
  CRF data
Investigtor´s MSS ratings [score points] at V5 | Day 57
  CRF data
Investigtor´s MSS ratings [score points] at V6 | Day 85
  CRF data
Investigtor´s MSS ratings [score points] at V7 | Day 141
  CRF data
Responders based on investigators´ ratings at V2, V3, V4, V5, V6 and V7 | 20 weeks
Responders based on patients´ ratings at V2, V3, V4, V5, V6 and V7 | 20 weeks

OTHER OUTCOMES:
CRS-related absenteeism from work | 20 weeks
  CRF data

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, Prof. Dr., Principal Investigator — Ghent University Hospital; Ear, Nose, Throat Medicine, Head & Neck Surgery; Upper Airway Research Laboratory - UZ Gent; De Pintelaan 185 / 1P1; 9000 Gent; Belgium.
Locations (1):
- Claus Bachert, Prof. Dr., Ghent, Belgium